CLINICAL TRIAL: NCT02483962
Title: The Efficacy of Red Vine Leaf Extract, Butcher's Broom, Horse Chestnut and Vitamin B6 in the Treatment of Symptoms Associated With Chronic Venous Insufficiency
Brief Title: Venavine Intensive® in the Treatment of Symptoms Associated With Chronic Venous Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FayroozKarriem200800851
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Venous Insufficiency
Keywords: Chronic
MeSH Terms: conditions — Venous Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelatine capsule (Placebo Comparator): Gelatine capsules containing no active ingredients, will be taken once per day, in the morning after breakfast, for 30 days. These capsules will be of identical appearance to the experimental comparator.
  Interventions: Other: Gelatine capsule
- Venavine Intensive® (Experimental): Gelatine capsules containing the active ingredients of: 360 mg red vine leaf extract, 60 mg of horse chestnut extract, 35 mg of butcher's broom extract and 3,2 mg of vitamin B6, will be taken once per day, in the morning after breakfast, for 30 days.
  Interventions: Other: Venavine Intensive®

INTERVENTIONS:
Other: Gelatine capsule — Gelatine capsules containing no active ingredients.
  Arms: Gelatine capsule
Other: Venavine Intensive® — Gelatine capsules containing 360 mg red vine leaf extract, 60 mg of horse chestnut extract, 35 mg of butchers broom extract and 3,2 mg of vitamin B6.
  Arms: Venavine Intensive®

SUMMARY:
Chronic Venous Insufficiency (CVI) occurs when the veins in the lower limbs can no longer sufficiently pump enough blood back to the heart. Symptoms may include: dull aching, cramping, itching or tingling in the calves, swelling, redness or any colour changes as well as thickening of the skin in the lower limbs. The most common indication of CVI is dilated veins known as varicose veins. CVI is a disorder found more commonly in females. Conventional treatments for CVI include vein ligation or stripping, elastic compression, valve reconstruction and sclerotherapy venous bypass. Amongst other treatment, exercise has also proven to be effective in improving CVI as it increases circulation, by increasing blood returning to the heart. A variety of herbal supplements have been proven to be safe and effective in the treatment of CVI. Red vine leaf extract has also been proven to be useful in the treatment of CVI. Previous studies on the red vine leaf extract have shown that it is an effective and safe treatment of CVI. Studies done on horse chestnut extract have stated that the extract increases venous tone and decreases capillary permeability. Butcher's broom extract has been proven to be effective in the treatment of CVI. There are currently no studies done on the combination of red vine leaf extract, butcher's broom extract, horse chestnut extract and vitamin B6.

The aim of this study is to determine the efficacy of a combination of red vine leaf extract (360mg), horse chestnut extract (60mg), butcher's broom extract (35mg) and pyridoxine (vitamin B6) (3.2mg) in the treatment of symptoms associated with CVI, using a Venous Clinical Severity Score questionnaire (VCSS) .

DETAILED DESCRIPTION:
This study is a 90 day, match paired, double-blinded, placebo-controlled study involving forty females participants between the ages of 30 and 55. Participants will be recruited via advertisements placed at the University of Johannesburg (UJ) Health Centre and on the campus. This sample group will be shared with another Homoeopathy Masters student, Xoliswa Mazibuko, who will be evaluating the changes in the quality of life using combination of red vine leaf extract, butcher's broom, horse chestnut extract and vitamin B6.

All consultations will take place at the UJ Health Centre, Doornfontein campus. The initial consultation will consist of signing of the Participant Information and Consent form as well as a Photograph Consent Form, followed by a screening test to confirm if participants qualify to participate in the study. All symptoms will be evaluated according to the Venous Clinical Severity Score (VCSS) questionnaire. Photographs of physical symptoms will also be taken, with the consent of the participant, in the initial consultation. Participants will be matched according to their age and severity of their symptoms. The bottles containing the placebo capsules will be placed in one box and the bottles containing the experimental capsules will be placed in another box. The boxes will be labelled X and Y. Each bottle will contain either 30 placebo capsules or 30 experimental capsules, as per their box group. The participants will then select a bottle from one of the boxes , thereby allocating themselves to either the experimental group or the control group. The participants will be requested to ingest one capsule from their selected bottle, every morning after breakfast for 30 consecutive days.

Follow up consultations will take place on days thirty, sixty and ninety. At each follow up consultation, the participants will be asked to complete the VCSS questionnaire, with the help of the researcher, and photographs of the same anatomical landmarks as taken in the initial consultation, will be taken. All photographs will be analysed by the Digimizer programme, which will calculate any changes in surface area from week one to week twelve. Photographs will be taken in such a way that the dignity and privacy of the participant is maintained.

Participants will be given medication for the next thirty days at each follow-up consultation excluding the final consultation (day 90).

If any other treatment or intervention is used during the duration of the study, they will be requested to notify the researcher.

Data will be collected from the questionnaire and analysed statistically with the assistance of a statistician at Statkon. Differences between the Inter-group will be analysed using the Friedman test with Wilcoxon post hoc test. To compare the different sets of data between the Intra-group, the Mann-Whitney test will be used. All photographs will be analysed by Digimizer programme.

ELIGIBILITY:
Inclusion Criteria:

* Females;
* aged 30 to 55 years;
* experiences at least three symptoms from Clinical, Etiologic, Anatomic, and Pathophysiologic (CEAP) C1-C4 of CVI which include varicose veins, tired or heavy legs, pain in the legs, tingling calves, venous oedema, induration of the legs, brown discolouration in the legs, skin changes such as erythema in the legs; and
* symptoms must be aggravated by walking/standing and symptoms are ameliorated by rest and limb elevation.

Exclusion Criteria:

* Pregnant or lactating females;
* taking chronic medication for cardiovascular disorder;
* have any chronic diseases that are not sufficiently managed;
* experiencing symptoms from CEAP C5-C6 of CVI, which includes venous ulceration;
* have a previous history of deep vein thrombosis;
* are on Warfarin or blood thinning medication;
* have any liver or kidney pathologies;
* are hypersensitive to any/all herbal extracts;
* are on any treatment (herbal or conventional) for CVI; and/or
* use compression stockings or Kinesio Taping therapy.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Severity of chronic venous insufficiency symptoms as measured by the Venous Clinical Severity Score (VCSS) | Every 30 days in a period of 90 days
  The VCSS is an effective tool in grading the severity of the symptoms of chronic venous insufficiency in response to treatment.

SECONDARY OUTCOMES:
Changes in surface area of the affected skin of the lower limbs as measured by photographs analysed by the Digimizer programme | Every 30 days in a period of 90 days
  The Digimizer programme calculates any changes in the surface area of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Razlog, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No